CLINICAL TRIAL: NCT05848947
Title: Study to Calculate the Radiation-Absorbed Dose of Technetium-99m Macroaggregated Albumin (99mTc-MAA) to the Whole Body and Non-Liver Critical Organs
Brief Title: SIR-Spheres Study to Calculate the Radiation-Absorbed Dose of 99mTc-MAA
Acronym: MAApping
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sirtex Medical (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STX2301
Record Dates: First submitted 2023-04-21; First posted 2023-05-08 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma; Carcinoma, Hepatocellular; Liver Neoplasm
Keywords: Technetium-99m macroaggregated-albumin (99mTc-MAA); SIR-Spheres Y90 resin microspheres treatment
MeSH Terms: conditions — Carcinoma; Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Technetium Tc 99m Aggregated Albumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 99mTc-MAA Injection (Other): Patients enrolled in the study will have 3 imaging scans taken after 99mTc-MAA Injection with the final scan occurring 18-24 hours after injection.
  Interventions: Drug: 99mTc-Macro Albumin Aggregate

INTERVENTIONS:
Drug: 99mTc-Macro Albumin Aggregate — Technetium-99m macroaggregated-albumin consists of macroaggregated-albumin particles labeled with technetium-99m (99mTc), with a size between 10 and 90 microns in diameter. 99mTc is a gamma emitting radioactive isotope commonly used for diagnostic localization studies.

SUMMARY:
The goal of this interventional clinical trial is to evaluate the dose of radiation of Technetium-99m macroaggregated-albumin (99mTc-MAA) after an intra-arterial injection to the whole body and non-liver critical organs in patients who are undergoing evaluation for SIR-Spheres treatment for hepatocellular carcinoma.

DETAILED DESCRIPTION:
The investigation is a prospective, single center, open label, single-arm study. Patients enrolled in the study will have 3 imaging scans taken after 99mTc-MAA injection, the final of which will occur between 18 and 24 hours post-injection.

ELIGIBILITY:
Inclusion Criteria:

1. Willing, able, and mentally competent to provide written informed consent
2. Age 18 or older at the time of consent
3. Patients who are being evaluated for SIR-Spheres treatment eligibility

Exclusion Criteria:

1. Patients who are contraindicated for SIR-Spheres treatment
2. Patients who are contraindicated for 99mTc-MAA per the manufacturer's package insert

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Murrey, MD, Principal Investigator — Inland Imaging
Locations (1):
- Inland Imaging, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gates VL, Singh N, Lewandowski RJ, Spies S, Salem R. Intraarterial Hepatic SPECT/CT Imaging Using 99mTc-Macroaggregated Albumin in Preparation for Radioembolization. J Nucl Med. 2015 Aug;56(8):1157-62. doi: 10.2967/jnumed.114.153346. Epub 2015 Jun 18. PMID 26089551
- [Background] Kappadath SC, Lopez BP. Organ-level internal dosimetry for intra-hepatic-arterial administration of 99m Tc-macroaggregated albumin. Med Phys. 2022 Aug;49(8):5504-5512. doi: 10.1002/mp.15726. Epub 2022 Jun 6. PMID 35612924
- [Background] McCollough CH, Bushberg JT, Fletcher JG, Eckel LJ. Answers to Common Questions About the Use and Safety of CT Scans. Mayo Clin Proc. 2015 Oct;90(10):1380-92. doi: 10.1016/j.mayocp.2015.07.011. PMID 26434964

RESULTS

PARTICIPANT FLOW:
Groups:
- 99mTc-MAA Injection: Patients enrolled in the study had 3 imaging scans taken after 99mTc-MAA Injection with the final scan occurring 18-24 hours after injection.
  99mTc-Macro Albumin Aggregate: Technetium-99m macroaggregated-albumin consists of macroaggregated-albumin particles labeled with technetium-99m (99mTc), with a size between 10 and 90 microns in diameter. 99mTc is a gamma emitting radioactive isotope commonly used for diagnostic localization studies.
Period: Overall Study
Arm/Group | 99mTc-MAA Injection
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 99mTc-MAA Injection
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Absorbed Dose (Gy) for the Whole Body
Time Frame: 18-24 hours
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | 99mTc-MAA Injection
Number analyzed (Participants) | 5
mGy | 0.941 (0.926)

2. Primary Outcome: Mean Absorbed Dose (Gy) for Critical Non-liver Organs
Time Frame: 18-24 hours
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | 99mTc-MAA Injection
Number analyzed (Participants) | 5
mGy
  Adrenal glands | 1.415 (1.524)
  Gallbladder | 4.855 (5.444)
  Heart | 0.736 (0.692)
  Kidney | 2.073 (3.401)
  Lungs | 1.701 (1.869)
  Pancreas | 1.221 (0.990)
  Spleen | 0.784 (1.037)
  Stomach | 2.530 (2.634)
  Upper bowel | 0.809 (0.785)

3. Primary Outcome: Mean Activity (Bq) for the Whole Body
Time Frame: 18-24 hours
Measure: Mean (Standard Deviation); unit: GBq
Arm/Group | 99mTc-MAA Injection
Number analyzed (Participants) | 5
GBq | 0.150 (0.014)

4. Primary Outcome: Mean Activity (Bq) for Critical Non-liver Organs
Time Frame: 18-24 hours
Measure: Mean (Standard Deviation); unit: GBq
Arm/Group | 99mTc-MAA Injection
Number analyzed (Participants) | 5
GBq
  Adrenal glands | 0.150 (0.014)
  Gallbladder | 0.148 (0.016)
  Heart | 0.150 (0.014)
  Kidney | 0.150 (0.014)
  Lungs | 0.150 (0.014)
  Pancreas | 0.150 (0.014)
  Spleen | 0.145 (0.018)
  Stomach | 0.150 (0.014)
  Upper bowel | 0.150 (0.014)

5. Primary Outcome: Effective Dose (Gy) for the Whole Body
Time Frame: 18-24 hours
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | 99mTc-MAA Injection
Number analyzed (Participants) | 5
mGy | 0.6 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the procedure until 18-24 hours post-procedure.
Arm/Group | 99mTc-MAA Injection
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon completion of the Study, Institution and Investigator may publish or present the Study Data subject to the following terms: a copy of any proposed publication or disclosure of the results of the Study will be given to the Sponsor for review at least thirty (30) days prior to the date of submission for publication (including abstracts) or of public disclosure.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT05848947/Prot_SAP_000.pdf